CLINICAL TRIAL: NCT03658395
Title: Randomized Trial of Laparoscopic Sacrocolpopexy With Posterior Repair to Reduce Obstructed Defecation Symptoms
Brief Title: Sacrocolpopexy With Posterior Repair Obstructed Defecation Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9457
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Vaginal Prolapse
Keywords: Vaginal, Prolapse, laparoscopic, sacrocolpopexy
MeSH Terms: conditions — Uterine Prolapse; Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LSCP Only (Active Comparator): A Y-shaped polypropylene mesh graft, 10 cm in standard length and tailored to each patient's anatomic specifications during surgery, is used utilizing robot-assisted Laparoscopic Sacrocolopopexy.
  Interventions: Procedure: Laparoscopic Sacrocolopopexy
- LSCP + PR (Active Comparator): The Laparoscopic Sacrocolopopexy involves a Y-shaped polypropylene mesh graft, 10 cm in standard length and tailored to each patient's anatomic specifications during surgery, utilizing robot-assisted Laparoscopic Sacrocolopopexy.
  In addition, patients will receive posterior repair. Posterior repair is performed by midline fascial plication. Plication of superficial perineal muscles (perineorrhaphy) is performed in conjunction with posterior repair. All repairs are performed using polydioxanone 2/0 for fascial repair and 4/0 polyglactin suture for skin closure.
  Interventions: Procedure: Laparoscopic Sacrocolopopexy; Procedure: Posterior repair

INTERVENTIONS:
Procedure: Laparoscopic Sacrocolopopexy — The LSCP surgery involves pulling up the bladder, vagina, and rectum using a Y-shaped mesh attached to the lower back bone
  Other Names: LSCP
Procedure: Posterior repair — The PR surgery involves tightening the tissue between the rectum and vagina to reduce vaginal bulging during bowel movements.
  Other Names: PR
  Arms: LSCP + PR

SUMMARY:
Participants who undergo laparoscopic sacrocolpopexy (LSCP) plus posterior repair (PR) will demonstrate greater improvement bowel symptom scores compared to participants who undergo LSCP alone at 3 months postoperatively.

DETAILED DESCRIPTION:
Those who provide informed consent will be randomized into either laparoscopic sacrocolpopexy (LSCP) alone or laparoscopic sacrocolpopexy (LSCP) plus posterior repair (PR). Participants will be randomized with equal probability to the LSCP only arm or LSCP plus PR arm.

The surgical technique for LSCP will be similar to that described by Paraiso et al. for LSCP [14] and by Elliott et al. for robot-assisted LSCP [15], with minor variations. A Y-shaped polypropylene mesh graft, 10 cm in standard length and tailored to each patient's anatomic specifications during surgery, will be used with all SCP procedures.

PR is performed by midline fascial plication. Plication of superficial perineal muscles (perineorrhaphy) is performed in conjunction with PR. All repairs are performed using polydioxanone 2/0 for fascial repair and 4/0 polyglactin suture for skin closure.

Participants will also complete questionnaires and undergo an endovaginal ultrasound (using a 9-16 MHz, 360° rotational transducer, type 8838, BK Medical, Peabody, MA) prior to surgery and three months following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female Gender
* Able to complete English language questionnaires
* Able to complete study visits for 6 months
* Bowel symptom score (PFDI-O) score ≥ 3
* Posterior vaginal bulge ≤2cm beyond the hymen

Exclusion Criteria:

* Age < 21
* Pregnancy
* History of colorectal surgery
* History of pelvic radiation
* Inflammatory bowel disease
* History of prior SCP

Ages: 21 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Primary Outcome (obstructed defecation symptoms) | 3 months postoperative
  The primary outcome of this study (AIM 1) is to compare bowel symptom scores in patients with ODS who undergo LSCP+PR compared to those who undergo LSCP only. Our primary outcome is a composite score from Questions 4, 7, and 8 of the PFDI-20.The responses to these three questions will be summed to a maximum score of 12. The ODS questionnaire is a validated, disease-specific, scoring system commonly used in the colorectal literature, which measures constipation severity, specifically outlet obstruction. Validated pelvic floor symptom survey data using the Pelvic Floor Distress Inventory-20 (PFDI-20), Pelvic Floor Impact Questionaire-7 (PFIQ-7), and Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire-12 (PISQ-12) will be obtained at study time points.

SECONDARY OUTCOMES:
Secondary Outcome (correlation between bowel symptoms scores and 3D ultrasound measurements) | 3 months postoperative
  For our secondary outcome, (AIM2) we will establish a correlation between bowel symptoms score and 3D ultrasound measurements of rectal support and LAM defects. Sonographic data will consist of Levator Ani Deficiency (LAD) score and Levator Plate Descent (LPDA) angle. Bowel symptom scores will be a subscale of the PFDI calculated using questions 4, 7, and 8 referring to splinting, straining, and incomplete emptying, respectively. The responses to these three questions will be summed to a maximum score of 12. We refer to these three questions collectively as the PFDI-Obstructed (PFDI-O), to represent obstructed defecation.

CONTACTS AND LOCATIONS:
Overall Officials: Lieschen Quiroz, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Frick AC, Paraiso MF. Laparoscopic management of incontinence and pelvic organ prolapse. Clin Obstet Gynecol. 2009 Sep;52(3):390-400. doi: 10.1097/GRF.0b013e3181b0bf69. PMID 19661755
- [Background] Elliott DS, Frank I, Dimarco DS, Chow GK. Gynecologic use of robotically assisted laparoscopy: Sacrocolpopexy for the treatment of high-grade vaginal vault prolapse. Am J Surg. 2004 Oct;188(4A Suppl):52S-56S. doi: 10.1016/j.amjsurg.2004.08.022. PMID 15476652